CLINICAL TRIAL: NCT00227916
Title: Motivational Interviews for Incarcerated Teens
Brief Title: Motivational Interviews for Incarcerated Teens - 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Lynda Stein, Professor, University of Rhode Island, National Institute on Drug Abuse (NIDA)
Purpose: Treatment
Other Study IDs: NIDA-13375-1; R01DA013375 (NIH); R01-13375-1; NCT00249184 (obsolete NCT alias)
Record Dates: First submitted 2005-09-27; First posted 2005-09-28 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Alcoholic Intoxication; Marijuana Abuse
Keywords: alcohol, marijuana
MeSH Terms: conditions — Alcoholic Intoxication; Marijuana Abuse | interventions — Behavior Therapy

INTERVENTIONS:
Behavioral: Behavior Therapy

SUMMARY:
The purpose of this study is to test the efficacy of an individual motivational interview for reducing alcohol and marijuana-related harm as well as alcohol and marijuana use in incarcerated teens.

DETAILED DESCRIPTION:
The objective of this research is to investigate ways to enhance motivation for treatment and effectively reduce substance abuse among juvenile offenders. Motivational intervention (MI) as preparation for residential treatment and for persons (including teens) with little motivation to change has been effective in reducing substance abuse. Thus, MI designed for delinquent youths who are required to attend substance abuse treatment may prove efficacious.

In this proposed randomized trial, a one-way design (MI + Standard Care [SC] v. Attention Control [AC] + SC) will be used to determine whether MI enhances subsequent treatment participation and reduces substance-related problems post discharge in substance using, delinquent youths. Teens will also receive a booster session of MI or AC prior to discharge. Primary outcome variables include alcohol and marijuana use, as well as related behaviors (illegal activity, sex or injuries while drunk or high). It is hypothesized that in comparison to teens receiving AC, youths receiving MI will participate more (by therapist and teen ratings) in SC and will show the lowest levels of heavy substance use and related problems after discharge. It is hypothesized that these effects will be mediated by stage of change, drug effect expectancies and self-efficacy.

This study will extend previous research by evaluating the use of MI with substance abusing teens in a correctional facility, and by expanding outcome measures to include alcohol and marijuana-related risk behavior (such as injuries and illegal activity when drunk or high) in this population. The development of effective interventions for substance using juvenile offenders has the potential to reduce substance abuse and crime in this population.

ELIGIBILITY:
Inclusion Criteria:

Teens will be included if they meet any of the following criteria: 1) in the year prior to incarceration they used marijuana regularly (at least monthly); 2) in the year prior to incarceration they drank regularly (at least monthly) or binged (>=5 for boys; >=4 for girls) over any two week period or less; 3) they used marijuana or drank in the 4 weeks before the offense for which they were incarcerated; or 4) they used marijuana or drank in the 4 weeks before they were incarcerated.

Exclusion Criteria:

Those teens sentenced for less than 4 months or greater than 12 months will be excluded from participation. We estimate that during year 1 we will exclude an additional 25% of youths because they will have previously participated in the study, and at year 2 we anticipate excluding an additional 49% of youths based on prior participation in the study.

Ages: 14 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2000-11; Primary Completion 2004-05 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Drug and alcohol use | baseline, 3 month in facility, 3 month post facility

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Stein, Ph.D., Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

REFERENCES:
- [Result] Stein LA, Graham JR. Ability of substance abusers to escape detection on the Minnesota Multiphasic Personality Inventory-Adolescent (MMPI-A) in a juvenile correctional facility. Assessment. 2005 Mar;12(1):28-39. doi: 10.1177/1073191104270838. PMID 15695741